CLINICAL TRIAL: NCT02903953
Title: Clinical Research Outside of Teaching Hospitals : Current Situation in North-eastern France
Brief Title: Clinical Research Outside of Teaching Hospitals (RECHNONU)
Acronym: RECHNONU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-01Obs-CHRMT
Record Dates: First submitted 2016-08-26; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-08

CONDITIONS: Medical Staff, Hospital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The very most part of clinical research in France takes place in teaching hospitals. Advantages to develop it in others hospitals are numerous: access to innovative treatments, improvement of healthcare quality, hospitals' attractiveness, increased inclusion rates and reduced selection bias. The objectives of the study are to report the current situation of clinical research outside of teaching hospitals in France.

DETAILED DESCRIPTION:
The very most part of clinical research in France takes place in teaching hospitals. Advantages to develop it in others hospitals are numerous: access to innovative treatments, improvement of healthcare quality, hospitals' attractiveness, increased inclusion rates and reduced selection bias. The objective the study is report the current situation of clinical research outside of teaching hospitals in France.

A three-stage survey was conducted between January and October 2012 in non-teaching hospitals of North-eastern France. First questionnaires were sent to administrative and medical boards of all hospitals with more than 100 beds, then to head doctors of every department in hospitals with more than 300 beds and finally meetings were organized with clinical research actors of 20 selected hospitals.

ELIGIBILITY:
Inclusion Criteria:

* non-teaching hospitals
* established in north-eastern France

Exclusion Criteria:

* more than 100 beds
* for the second stage only:
* less than 300 beds

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-teaching hospitals of North-eastern France
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Description of the clinical research in non-teaching hospitals of north-eastern France | 1 year
  Self-Assessment Questionnaire

SECONDARY OUTCOMES:
Specificities of each centers in clinical research | 1 year
  Self-Assessment Questionnaire
Problems to solve for developing clinical research | 1 year
  semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Christophe GOETZ, MD, Study Director — CHR Metz-Thionville

IPD SHARING:
Plan to Share IPD: No